CLINICAL TRIAL: NCT01256216
Title: A Comparison of Signature Custom Cutting Guides and Computer Assisted Surgery Techniques With the Vanguard Knee System
Brief Title: Signature Versus Computer Assisted Surgery Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 121509
Record Dates: First submitted 2010-05-12; First posted 2010-12-08 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Joint Disease
Keywords: Arthritis; Osteoarthritis; Arthroplasty
MeSH Terms: conditions — Joint Diseases; Arthritis; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Signature Custom Cutting Guides (Other): Patients receiving a Vanguard Total Knee implanted utilizing non implantable Signature Cutting Guides Surgical Technique.
  Interventions: Device: Total Knee Replacement with Vanguard Total Knee
- CAS (Computer Assisted Surgery) (Other): Patients receiving a Vanguard Total Knee implanted utilizing non implantable Computer Assisted Surgery Technique.
  Interventions: Device: Total Knee Replacement with Vanguard Total Knee

INTERVENTIONS:
Device: Total Knee Replacement with Vanguard Total Knee — Patients indicated for a total knee replacement utilizing the Vanguard Total Knee System.

SUMMARY:
The purpose of the data collection is to document the performance and clinical outcomes of the Vanguard Knee using Signature Custom Cutting Guides and Computer Assisted Surgery.

DETAILED DESCRIPTION:
The purpose of this prospective clinical data-collection is to document the performance and clinical outcomes of the Vanguard® Knee System using Signature™ Custom Guides and Computer Assisted Surgery.

FDA has cleared the Vanguard Knee via premarket notification 510(k) K023546, K033489, and K050222. FDA has cleared the software for the Signature™ Custom Guides via premarket notification 510(k) K073449. The data gathered will be collated and used to provide feedback to design engineers, support marketing efforts, answer potential questions from reimbursement agencies, and will serve as a part of Biomet's Post Market Surveillance System.

Function will be assessed through the Knee Society Score. Survivorship will be documented by asking the surgeon to document revisions and complications.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are identical to the indications for use stated in the FDA cleared labeling for the device (510(k) K023546, K033489, and K050222).

These indications are stated below:

* Painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more compartments are involved.
* Correction of varus, valgus, or posttraumatic deformity.
* Correction or revision of unsuccessful osteotomy, arthrodesis, or failure of previous joint replacement procedure.
* The Regenerex™ femoral augments are indicated for use with the Vanguard® Total Knee System.
* The Regenerex™ tibial augments are indicated for use with standard and offset Biomet® Tibial Trays.

Patient selection factors to be considered include:

* Need to obtain pain relief and improve function
* Ability and willingness of the patient to follow instructions, including control of weight and activity level
* A good nutritional state of the patient, and
* The patient must have reached full skeletal maturity
* Femoral components and tibial tray components with porous coatings are indicated for cemented and uncemented biological fixation application. Non-coated (Interlok™) devices and all polyethylene patellar components are indicated for cemented application only.

Exclusion Criteria: Exclusion criteria are identical to the contraindications stated in the FDA cleared labeling for the device 510(k) K023546, K033489, and K050222. These contraindications are stated below:

* Absolute contraindications include: infection, sepsis, and osteomyelitis
* Relative contraindications include:
* Uncooperative patient or patient with neurologic disorders who is incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair bone formation,
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, neuromuscular disease
* Incomplete or deficient soft tissue surrounding the knee.
* Biomet® Microplasty™ Tibial Trays are contraindicated for use with constrained bearings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Mechanical Alignment | Data Collected at 0-10 Weeks; but Analyzed at Completion of Study
  Angle between femoral head, center of knee, and talus.

SECONDARY OUTCOMES:
Knee Society Objective Score | Completion of Study
  Objective Scoring of Knee Society score is the clinical assessment which includes the sum of range of motion, stability, flexion contracture, extension lag, and alignment scores.

CONTACTS AND LOCATIONS:
Overall Officials: Russell A Schenck, PhD, Study Director — Zimmer Biomet
Locations (1):
- Russells Hall Hospital, Dudley, United Kingdom